CLINICAL TRIAL: NCT02107391
Title: Randomized, Open-label, Parallel-group, Multi-centre Phase II Clinical Trial of Active Cellular Immunotherapy With Preparation DCVAC/PCa in Combination With Hormone Therapy in Patients With Metastatic Prostate Cancer
Brief Title: Phase II Study of DCVAC/PCa Added to Hormone Therapy for Men With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP002; 2011-004986-34 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2015-06

CONDITIONS: Prostate Cancer
Keywords: Immunotherapy; Prostate Cancer; Biological; Vaccine; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DCVAC/PCA added Standard Hormone Therapy (Experimental): Combination therapy with Dendritic Cells DCVAC/PCa added on to a Standard of Care Hormone Therapy
  Interventions: Biological: Dendritic Cells DCVAC/PCa
- Standard of Care Hormone Therapy (Active Comparator): Standard of Care Hormone Therapy as an Active Comparator Goserelin Acetate Leuprolide Acetate
  Interventions: Drug: Leuprolide acetate; Drug: Goserelin Acetate

INTERVENTIONS:
Biological: Dendritic Cells DCVAC/PCa — Combination therapy with DCVAC/PCA add on to and Standard of Care Hormone Therapy
  Arms: DCVAC/PCA added Standard Hormone Therapy
Drug: Leuprolide acetate — Standard of Care Hormone Therapy as an Active Comparator
  Other Names: Lupron
  Arms: Standard of Care Hormone Therapy
Drug: Goserelin Acetate — Standard of Care Hormone Therapy as an Active Comparator
  Other Names: Zoladex
  Arms: Standard of Care Hormone Therapy

SUMMARY:
The purpose of this study is to determine whether DCVAC/PCa added onto hormone therapy can improve PSA progression times for patients with Metastatic Prostate Cancer.

DETAILED DESCRIPTION:
Use of vaccine to improve Prostate Specific Antigen (PSA) levels.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years and older
* Histologically confirmed prostate adenocarcinoma
* Presence of bone or soft tissue metastasis (by CT or PET or MRI and/or scintigraphy)
* Androgen deprivation therapy using Luteinizing-hormone-releasing hormone ( LHRH) analogues commenced at least one month and at most three months prior randomization or orchiectomy performed at least one month and at most three months prior randomization
* Serum testosterone level at screening (≤ 1.7 nmol/l, resp. ≤ 50 ng/dL)
* Eastern Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

* Confirmed brain and/or leptomeningeal metastases
* Prior or ongoing chemotherapy for prostate cancer
* Peripheral neuropathy of Common Toxicity Criteria (CTC) grade 2 or greater
* Other uncontrolled intercurrent illness
* Treatment with immunotherapy against prostate cancer
* Clinically significant cardiovascular disease
* Active autoimmune disease requiring treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with PSA Progression | 104 weeks

SECONDARY OUTCOMES:
Proportion of patients with Progression of Disease | 0, 6, 16, 28, 40, 52, 65, 78, 91, 104 weeks
Frequency of Adverse Events | 0, 2, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 52, 65, 78, 91, 104 weeks
Frequency of Skeletal Related Events | 0, 2, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 52, 65, 78, 91, 104 weeks
Changes in Quality of Life (QOL) assessed by EORTC QLQ-C30 | 0, 16, 28, 40, 52, 52, 65, 78, 91, 104 weeks
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) form C30
Changes in Pain assessed by EORTC QLQ-C30 | 0, 16, 28, 40, 52, 52, 65, 78, 91, 104 weeks
  Pain Scale from European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) form C30

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Scheiner, PhD, Study Director — Sotio-Accord
Locations (9):
- Czechia (9):
  - Jablonec nad Nisou
  - Jihlava
  - Liberec
  - Mníšek pod Brdy
  - Olomouc
  - Pilsen
  - Prague
  - Ústí nad Labem
  - Zlín